CLINICAL TRIAL: NCT05971849
Title: Dampening the Reproductive Axis With Continuous Kisspeptin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stephanie B. Seminara, MD (Other)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023P001356
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Reproductive Disorder; PCOS; Polycystic Ovary Syndrome
Keywords: reproductive disorders; kisspeptin; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- kisspeptin (Experimental): IV administration of kisspeptin 112-121; 24-hour infusion, up to 2 boluses.
  Interventions: Drug: kisspeptin 112-121

INTERVENTIONS:
Drug: kisspeptin 112-121 — IV infusion of kisspeptin 112-121 x 24 hours; up to two IV boluses of kisspeptin
  Other Names: metastin 45-54

SUMMARY:
The goal of this study is to assess response to kisspeptin as well as the baseline patterns of luteinizing hormone (LH) secretion in individuals with polycystic ovarian syndrome (PCOS).

DETAILED DESCRIPTION:
Assignment: All study subjects will undergo the same interventions. Baseline LH secretion patterns of individuals with PCOS will be compared to their LH secretion patterns while receiving a kisspeptin infusion.

Delivery of Interventions:

* Prior to the inpatient study visit, the subjects will undergo a review of their medical history, physical exam, and screening laboratories.
* On the day of the study, the subjects will have an intravenous (IV) line placed and

  * Undergo up to q10 min blood sampling x 36 hours
  * Receive an infusion of kisspeptin x 24 hours
  * Receive up to two kisspeptin IV boluses

ELIGIBILITY:
* Ages 18-45 years
* A history of clinical diagnosis of PCOS or equivalent clinical features
* BMI >18.5 and <35 kg/m2
* Normal blood pressure (systolic BP < 140 mm Hg, diastolic > 90 mm Hg)
* Laboratory studies:

  * Negative human chorionic gonadotropin (hCG) pregnancy test prior to kisspeptin administration
  * Hemoglobin no less than 0.5 g/dL below the lower limit of the reference range for healthy women
* Not using hormonal medication or willing to complete an appropriate washout for that particular medication and its method of administration
* No current or recent use of a medication that, in the opinion of a study investigator, can modulate the reproductive axis or willing to complete an appropriate washout for that particular medication and its method of administration
* No excessive alcohol consumption (>10 drinks/week) and/or ongoing use of illicit drugs

  • Any current use of marijuana will be evaluated by a study medical professional to determine if it is expected to impact study participation
* Not pregnant or trying to become pregnant
* Not breastfeeding
* No history of bilateral oophorectomy (both ovaries removed)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-04-27 (Actual)

PRIMARY OUTCOMES:
Average change in LH pulse frequency | 6 hours prior to kisspeptin infusion compared to the final 6 hours of kisspeptin infusion
  Average change in LH pulse frequency before and during kisspeptin infusion
Average change in LH pulse amplitude | 6 hours prior to kisspeptin infusion compared to the final 6 hours of kisspeptin infusion
  Average change in LH pulse amplitude before and during kisspeptin infusion

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No